CLINICAL TRIAL: NCT05537246
Title: The Importance of Preoperative Arterial Stiffness Measurement in Predicting Hemodynamic Changes in Hypertensive and Normotensive Patients Undergoing Spinal Anaesthesia
Brief Title: The Relationship Between Arterial Stiffness and Hemodynamic Responses in Patients With Spinal Anesthesia
Acronym: SpiASHT
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Associate Professor, Aydin Adnan Menderes University
Other Study IDs: SpiASHT
Record Dates: First submitted 2022-07-26; First posted 2022-09-13 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Arterial Stiffness; Hypertension; Spinal Anaesthesia
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP HT: In the preoperative evaluation, after arterial blood pressure measurement was made 3 times; Hypertension group was defined as the patients who did not use drugs that are effective on the cardiovascular system, whose SBP value was higher than 140 mmHg, or those who were diagnosed with hypertension and were using drugs with a SBP value higher than 140 mmHg.
  Interventions: Procedure: PWV
- GROUP NORMO: As a result of 3 measurements and medical histories of the cases, those who did not use drugs effective on the cardiovascular system and whose SBP value was lower than 140 mmHg were called the normotensive group.
  Interventions: Procedure: PWV

INTERVENTIONS:
Procedure: PWV — All cases were evaluated in the service before surgery. Pulse wave velocity measurement was performed with the MOBİL-O-GRAPH device, which is one of the noninvasive methods. Before measuring from patients; It was confirmed that there was no coffee/cigarette consumption within 30 minutes. After resting for 5 minutes in a quiet room, the cuff of the appropriate size was tied to the arm in such a way that it came to the brachial artery. The data recorded by the tonometer was transferred to the computer program. Care was taken that the patient did not move or talk during the measurement.

SUMMARY:
The aim of this study is to investigate the importance of pulse wave velocity, an indicator of arterial stiffness, in predicting hemodynamic changes in normotensive and hypertensive patients undergoing spinal anesthesia.

DETAILED DESCRIPTION:
The prospective cross-sectional study will be carried out between September 1, 2021 and September 1, 2022 at Aydin Adnan Menderes University Faculty of Medicine. Patients aged eighteen and over who will undergo lower extremity surgery under spinal anesthesia will be included in the study.

During the preoperative evaluation, the patient will be asked about age, weight, height, smoking and alcohol use history. At the same time, hypertension disease (if any, drugs used), diabetes (if any, drugs used), hyperlipidemia (if any, drugs used) and other diseases and drugs used will be recorded.

Before surgery, hemodynamic data (systolic arterial blood pressure, diastolic arterial blood pressure, mean arterial blood pressure, heart rate and oxygen saturation), arterial stiffness measurement (pulse wave velocity) will be evaluated in the patient preparation room. Arterial stiffness measurement will be made with the oscillometric mobil-o-graph device in the anesthesia department.

Hemodynamic data is recorded by the anesthesia device 1.,3.,5.,10.,20. minutes during surgery. Intraoperative hypotension is accepted as a 20% reduction in systolic arterial blood pressure evaluated before anesthesia. Using this data recorded on the monitor, reductions of 20% or more in systolic arterial blood pressure will be recorded as hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective lower extremity surgery
* 18 years and over
* who agreed to participate in the study
* ASA I-II

Exclusion Criteria:

* Undergoing cardiovascular or neurological surgery within 6 months
* Unwilling to participate in the study
* Undergoing prosthetic valve surgery
* Vasculitis
* Peripheral artery disease
* Under the age of 18
* Conditions in which spinal anesthesia is contraindicated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-II patients who will undergo elective lower extremity surgery under spinal anesthesia in the orthopedic operating room were selected.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Arterial blood pressure | 1., 3., 5., 10., 20. minute
  After spinal anesthesia, SBP, DBP, MAP, HR and SpO₂ values of all patients were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Yılmaz, Principal Investigator — institutional affiliation
Locations (2):
- Turkey (Türkiye) (2):
  - Sinan Yılmaz, Efeler, Aydın
  - Aydin Adnan Menderes University Faculty of Medicine, Department of Anesthesiology and Reanimation, Aydin

IPD SHARING:
Plan to Share IPD: No